CLINICAL TRIAL: NCT05259566
Title: Evaluating the Potential Impact of a Menthol Ban in Cigarettes and E-cigarettes Among Current Menthol Smokers
Brief Title: Potential Impact of Menthol Ban in Cigarettes and E-cigarettes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000032211; 1R01DA054993-01A1 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Smoking
Keywords: menthol; E-cigarette; cigarette
MeSH Terms: conditions — Tobacco Smoking; Vaping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no menthol ban (No Intervention): usual menthol cigarettes and menthol flavored e-cigarette available
- menthol ban in cigarettes only (Experimental): non-menthol cigarettes and menthol flavored e-cigarette available
  Interventions: Behavioral: menthol ban in cigarettes only
- menthol ban in both cigarettes and e-cigarettes (Experimental): non-menthol cigarettes and tobacco flavored e-cigarette available,
  Interventions: Behavioral: total menthol ban

INTERVENTIONS:
Behavioral: menthol ban in cigarettes only — menthol ban in cigarettes only, menthol available in e-cigarette
  Arms: menthol ban in cigarettes only
Behavioral: total menthol ban — menthol ban in both cigarettes and e-cigarettes
  Arms: menthol ban in both cigarettes and e-cigarettes

SUMMARY:
Menthol cigarette use remains a major public health problem and the FDA has proposed to ban menthol in cigarettes. However, additional evidence is needed to understand whether menthol flavor in e-cigarettes is important for harm reduction among menthol cigarette smokers in the context of a menthol cigarette ban. The primary aim of this project is to understand how the availability of menthol vs tobacco flavor e-cigarettes influences switching and reduces smoking behavior among adults who currently smoke menthol cigarettes to understand the potential effects in the context of a ban of menthol cigarettes.

DETAILED DESCRIPTION:
Menthol cigarette use remains a major public health problem and the FDA has proposed to ban menthol in cigarettes. However, additional evidence is needed to understand whether menthol flavor in e-cigarettes is important for harm reduction among menthol cigarette smokers in the context of a menthol cigarette ban.

The primary aim of this project is to understand how the availability of menthol vs tobacco flavor e-cigarettes influences switching and reduces smoking behavior among adults who currently smoke menthol cigarettes to understand the potential effects in the context of a ban of menthol cigarettes. The secondary aim of this project is to understand whether smoking behavior outcomes differ by race to understand the impact of these potential menthol ban policies on addressing tobacco-related health disparities.

This single site study will take place over a 4 year study period; approximately 14 weeks for each participant's completion.

150 adults who currently smoke menthol cigarettes will be enrolled and prospectively randomized using a randomization ratio of 1:1:1 to 1 of 3 groups (N=50 per group). Following an initial baseline period where participants have access to their usual menthol cigarettes (Phase I), participants will receive tobacco products to use for 8 weeks based on their assigned group modeling 3 possible regulatory scenarios (Phase II): 1) no menthol ban (menthol cigarettes and e-cigarettes available), 2) menthol ban in cigarettes only (non-menthol cigarettes and menthol e-cigarettes available), 3) menthol ban in both cigarettes and e-cigarettes (non-menthol cigarettes and tobacco e-cigarettes available). A follow-up survey at week 12 will assess tobacco use outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Age 21 or older
* Able to read English
* Currently smoking cigarettes
* Willing to try e-cigarettes
* In good general health

Exclusion Criteria:

* Seeking smoking cessation treatment
* Serious psychiatric or medical condition
* Use of other drugs
* Unable or unwilling to complete study protocol
* Contraindications for study procedures based on medical history

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Average number of cigarettes smoked per day in the past week to evaluate changes in smoking behavior | From Week 0 to week 8
  Participants will report the total number of cigarettes consumed each day using the well-validated timeline follow-back (TLFB) interview methods to assess change.

SECONDARY OUTCOMES:
Percent days smoke-free | From Week 0 to week 8
  Participants will report the number of smoke free days over the 8 week study period. Percent days smoke-free will be determined using the TLFB interview methods.
Changes in nicotine dependence using the Nicotine Dependence for Daily Smokers Scale | From Week 0 to week 8
  Changes in nicotine dependence will be measured using the Nicotine Dependence for Daily Smokers Scale from the NIH Patient Reported Outcome Measure Information System (PROMIS) bank. Scores are averaged across 4 items, min=1, max=5. Higher scores indicate greater nicotine dependence.
Change in Quitting motivation and confidence | Week 0 and week 8
  Quitting motivation and confidence will be assessed using the PhenX Toolkit using the items "How motivated are you to quit smoking?" and "How confident are you that you could quit smoking if you tried?" rated from 1 (not at all) to 10 (extremely).
Quit intentions using the Stages of Change Assessment | Week 8
  Participants will report their plans to quit smoking in the next 30 days based on Stages of Change Assessment, on a scale from 0 (I have absolutely no intention of quitting smoking) to 10 (I have made a firm decision to quit in the next 30 days). Higher scores indicate the more intention to quit.

OTHER OUTCOMES:
Percent days of e-cigarette use | From Week 0 to week 8
  Participants will report the number of days using the e-cigarette over the 8 week study period using the TLFB interview
Number of quit attempts during follow-up | Week 12
  Number of quit attempts at the 12-week follow-up, measured by the TLFB interview methods.

CONTACTS AND LOCATIONS:
Overall Officials: Krysten Bold, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study data is collected and cleaned, and the primary paper is published, de-identified study data will be available for research purposes to qualified individuals within the scientific community by request from the PI or through the National Addiction & HIV Data Archive Program (NAHDAP) an NIH-funded repository, consistent with NIH guidelines for the timely release and sharing of resources. Additional data documentation and codebooks defining relevant variables, terminology, and scoring guidelines for scale scores will be deposited and made available for sharing along with de-identified data.
Supporting Information: Analytic Code
Time Frame: After the study data is collected and cleaned, and the primary paper is published, de-identified study data will be made available to individuals within the scientific community by request from the PI or through NIH data repository.
Access Criteria: As we plan to use NAHDAP, which is an NIH-funded repository, this repository has policies and procedures in place that will provide access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.

REFERENCES:
- [Derived] Bold KW, Sharma A, Haeny A, Gueorguieva R, Buta E, Baldassarri S, Lempert L, Krishnan-Sarin S, O'Malley S. A randomized controlled trial of potential tobacco policies prohibiting menthol flavor in cigarettes and e-cigarettes: a study protocol. BMC Psychiatry. 2024 Mar 12;24(1):201. doi: 10.1186/s12888-024-05619-0. PMID 38475757